CLINICAL TRIAL: NCT01099280
Title: Induction of Labor in Term Premature Rupture of Membranes: A Comparison Between Oxytocin and Dinoprostone Followed Six Hours Later by Oxytocin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: No sponsor, Bakırkoy Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Gungorduk-08
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2010-03

CONDITIONS: Labor; Induction; PROM (Pregnancy)
Keywords: induction of labor in term; premature rupture of membranes; dinoprostone; oxytocin
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

ARMS (2):
- oxytocin group (Experimental): 2 milliunits/min and doubled every 30 minutes to a maximum of 32 milliunits/min or until four contractions in 10 minutes was achieved
  Interventions: Drug: SYNPITAN FORT 5 IU
- dinoprostone and oxytocin (Experimental): a single dose sustained-released dinoprostone into the posterior vaginal fornix. A standard intravenous oxytocin was administered 6 hours after the insertion of the vaginal pessary. An initial dose of 2 mU/min was increased at 30 minute intervals by 2 mU/min to a maximum dose 32 mU/min or until four contractions in 10 minutes was achieved
  Interventions: Drug: Propess,SYNPITAN FORT

INTERVENTIONS:
Drug: SYNPITAN FORT 5 IU — A standard intravenous oxytocin was administered 6 hours after the insertion of the vaginal pessary. An initial dose of 2 mU/min was increased at 30 minute intervals by 2 mU/min to a maximum dose 32 mU/min or until four contractions in 10 minutes was achieved. Once started, oxytocin infusion was continued to delivery unless otherwise indicated. The pessary has been removed if it was still present 12 h after placement; or if worrisome FHR pattern persisted
  Arms: oxytocin group
Drug: Propess,SYNPITAN FORT — a single dose sustained-released dinoprostone into the posterior vaginal fornix. A standard intravenous oxytocin was administered 6 hours after the insertion of the vaginal pessary. An initial dose of 2 mU/min was increased at 30 minute intervals by 2 mU/min to a maximum dose 32 mU/min or until four contractions in 10 minutes was achieved
  Arms: dinoprostone and oxytocin

SUMMARY:
Prelabor rupture of membranes (PROM) is most commonly defined as rupture of membranes before the onset of labor and occurs in 8% of term pregnancies. A prolonged interval from rupture of membranes to delivery is associated with an increase in the incidence of chorioamnionitis and neonatal sepsis. The management of the term patients with PROM, especially those with an unfavorable cervix, remains controversial. Management options to choose from are immediate induction of labor versus delayed induction or expectant management. Several reports have detailed an increase in maternal and neonatal morbidity with expectant management, whereas active management leads to a shorter interval from PROM to delivery, reducing the risk of postnatal infections. In addition, active management is preferred by patients.

The investigators know that, neonatal intensive care admission, variable decelerations, and primary cesarean delivery rates are positively correlated with a longer admission-to-labor-onset interval in women with PROM . So, to reduce the induction to delivery times, concurrent oxytocin infusion with dinoprostone vaginal pessary use for labor induction in women with PROM may be beneficial. Several studies have shown shorter induction-to-delivery interval with concurrent oxytocin infusion with prostaglandin agent at initiation of labor . However, in these studies, there is a a paucity information in PROM labor induction. Only one randomized control trial have compared the efficacy of concurrent dinoprostone and oxytocin and oxytocin alone in women with term PROM . This study indicated that concurrent vaginal dinoprostone and intravenous oxytocin conferred no advantage over intravenous oxytocin alone for the outcomes of interest, including length of labor patient satisfaction or risk for cesarean delivery. Unfortunately, this study was limited by small sample size.

The aims of this randomized study was to compare two protocols (oxytocin vs. sustained-release dinoprostone followed six hours later by oxytocin) for induction of labour in women with PROM at term and an unfavorable cervix.

ELIGIBILITY:
Inclusion Criteria:

* Women with a live singleton fetus at term [37-42 weeks of gestation in cephalic presentation
* reactive nonstress test (NST)
* presenting with PROM
* a Bishop score of 5 or less before the onset of labor
* an absence of spontaneous contractions

Exclusion Criteria:

* Women in active labor
* previous uterine surgery,
* antepartum hemorrhage,
* chorioamnionitis,
* contraindication to prostaglandin use (bronchial asthma, glaucoma), *contraindication to vaginal delivery,
* multiple pregnancy,
* non-vertex presentation
* major fetal anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
the number (rate) of women who succeeded in delivering vaginally within 24 h of the initiation of the labor induction protocol | 24 hours

SECONDARY OUTCOMES:
labor induction-to-delivery interval | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Women and Children Hospital, Istanbul, Yanimahalle, Turkey (Türkiye)